CLINICAL TRIAL: NCT06604845
Title: A Single-blind Randomised Controlled Trial of Group Cognitive Behavioural Therapy (CBT) Versus Activity Group Control Condition for Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: A Comparison of Group Cognitive Behavioural Therapy (CBT) and Structured Activity Group for Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EPM Dnr 2024-02227-01; 2023-01505 (Other Grant/Funding Number: Forte)
Record Dates: First submitted 2024-09-17; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Attention Deficit Hyperactivity Disorder (ADHD); Cognitive Behavioral Therapy; Controlled Clinical Trials, Randomized; Adults
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group cognitive behavioural therapy (Experimental): Group CBT based on an adapted version of individual CBT for ADHD according to Safren's manual "CBT for ADHD/Mastering Your Adult ADHD".
  Interventions: Behavioral: Group cognitive behavioural therapy (CBT)
- Activity group (Active Comparator): The Activity group is a structured manualised group intervention designed by clinicians and researchers at Sahlgrenska University Hosptial.
  Interventions: Other: Activity group

INTERVENTIONS:
Behavioral: Group cognitive behavioural therapy (CBT) — CBT based on Safren's manual "CBT for ADHD/Mastering Your Adult ADHD"20 adapted for group format. The program includes psychoeducation and cognitive restructuring and aims to improve ADHD symptoms, especially planning, organisation, attention and adaptive thinking. The CBT groups will meet at the clinic weekly for 12 weeks for 2 hours including a break in the middle. The groups are led by two clinicians.
  Arms: Group cognitive behavioural therapy
Other: Activity group — The Activity group is a structured manualised group intervention designed for this and planned future studies of psychosocial treatments for adults with ADHD and/or autism. The program includes group discussions, peer-sharing and social every-day life activities. The Activity groups will meet at the clinic weekly for 12 weeks for 2 hours including a break in the middle. The groups are led by two trainers.
  Arms: Activity group

SUMMARY:
Many adults with attention deficit hyperactivity disorder (ADHD) experience difficulties with inattention, planning and impulsivity that impacts work and social life negatively also after treatment with medication. There are various psychological treatments aiming to improve these symptoms, but it is not known if they work or not.

The goal of this clinical trial is to evaluate group cognitive behavioural therapy (CBT) for adults with attention deficit hyperactivity disorder (ADHD) in comparison to an active control group consisting of a discussion and activity group. Previous research suggests that group CBT works about equally well as other structured group activities. The main questions the researchers aim to answer are if group CBT work better than activity groups to:

* Improve symptoms of ADHD
* Improve general mental health and life quality
* Improve every-day functioning

The researchers also want to learn if group CBT or activity groups work better for some people with ADHD depending on individual characteristics such as

• type of symptoms, age, gender or co-occurring psychiatric diagnoses.

The comparison is a manualised structured activity group given at the same number of sessions and same group size. All participants will visit our clinics at 12 occasions. They will:

* Fill in questionnaires before and after the group intervention, and online after 6 and 12 months
* Do cognitive testing before and after the intervention

DETAILED DESCRIPTION:
Despite medical treatment, many adults with ADHD experience residual symptoms that negatively affect work performance and social life. Hence, several psychological interventions targeting these symptoms have been developed, but the treatment effects are still unclear due to lack of controlled clinical trials.

In this single-blind randomised controlled clinical trial, we will evaluate the effects of group CBT based on Safren's manual "CBT for ADHD/Mastering Your Adult ADHD" (Safren SA et al, Behav Res Ther, 2005), compared to an active control group. The control intervention is a manualised activity group that contains the same non-specific therapeutic elements as the treatment but no active CBT components. For dose equivalence, activity groups will be given with the same same number and length of sessions, and the same frequency, as the treatment conditions. Since therapist experience is known to influence outcomes, the activity groups will be held by staff with equivalent training and experience to those giving the treatment groups.

Consenting patients assessed eligible for treatment will be randomly assigned to treatment or control group using a standard digital randomisation generator with an allocation of 1:1. Patients and clinicians rating outcomes will be blind to group assignment.

Pre- and post intervention, and at 6 months and 12 months follow-up, the patient's ADHD symptoms, symptoms of anxiety and depression and general functioning will be assessed by experienced clinicians and with validated self-rating scales. Treatment fidelity and expectation will be compared for the therapy and control groups and adverse events will be registered.

An exact power calculation for estimation of sample sizes cannot be performed since effect sizes are not known. Based on a previously published studies of Safren's CBT individually administered, and general consensus of what is a clinically meaningful improvement in psychological treatments for other psychiatric diagnoses, we expect that 60 patients per arm will be sufficient for detection of clinically relevant effect sizes of approximately Cohen's d 0.3-0.4. A statistician will make a blind Bayesian stop analysis (Svensson JE et al, J Cereb Blood Flow Metab, 2021) for every 20-25 patients, and based on the results we can decide to halt the study if sufficient power has been achieved earlier than after 60 patients. Full attrition analysis with intention to treat (ITT) analysis will be performed to investigate and minimize attrition bias.

ELIGIBILITY:
Inclusion Criteria: Fulfilling criteria for ADHD , motivation and practical possibility to participate in the treatment.

-

Exclusion Criteria: Ongoing psychosis or suicidality, severe self-injury, intellectual disability and insufficient Swedish language skills.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Adult ADHD Self-Report Scale (ASRS) | From enrollment to the follow-up 12 months after end of treatment
  ASRS is a self-reported symptom questionnaire for adults with ADHD. It has 18 questions about how often the participant experiences a certain symptom, with five response choices ranging from 0 (never) to 4 (very often) points.
Change in Clinical Global Impressions-Severity (CGI-S) | At enrollment and after 12 weeks at end of treatment
  CGI-S is a 7-point scale where the clinician rate the severity of the patients illness at the time of assessment.

SECONDARY OUTCOMES:
Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM) | From enrollment to the follow-up 12 months after end of treatment
  CORE-OM is a self-rating questionnaire covering general psychiatric symptoms, well-being and functioning. It has 34 questions about how often the participant experiences a certain symptom, with five response choices ranging from 0 (not at all) to 4 (most or all of the time) points.
Brunnsviken Brief Quality of Life Inventory (BBQ) | From enrollment to the follow-up 12 months after end of treatment
  BBQ is a validated brief version of the self-rating Quality of Life Scale, with higher sensitivity to change. It consists of 12 statements and the participant indicates how much they agree with each statement in five response choices ranging from 0 (do not agree at all) to 4 (agree completely).
Colour word Interference Test (CWIT) | At enrollment and after 12 weeks at end of treatment
  The cognitive task CWIT from the Delis-Kaplan Executive Function System (D-KEFS) is a version of the Stoop test aiming to measure switching and inhibition.
Trail Making Test (TMT) | At enrollment and after 12 weeks at end of treatment
  The cognitive test TMT from the Delis-Kaplan Executive Function System (D-KEFS) is used to measure processing speed and cognitive flexibility.

OTHER OUTCOMES:
Treatment Credibility questionnaire (TCS) | At enrollment and after 12 weeks at end of treatment
  Swedish version of the TCS (Borkovec TD et al, J Behav Ther Exp Psychiatry, 1972) for assessment of treatment fidelity and expectation in both participants with ADHD and clinicians administering the CBT and activity groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Sahgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
Most individual data will be part of patients medical records.